CLINICAL TRIAL: NCT07328451
Title: A Phase 1b, Multicenter, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DNL628 in Participants With Early Alzheimer's Disease
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DNL628 in Participants With Early Alzheimer's Disease
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: DNLI-K-0001; 2025-523515-11-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-24; First posted 2026-01-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease, Early Onset
Keywords: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor staff directly interacting with the site (clinical operations and medical monitor) will be blinded but may be unblinded if necessary to ensure participant safety.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental)
  Interventions: Drug: DNL628
- Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DNL628 — Multiple ascending doses
  Arms: Experimental Arm
Drug: Placebo — Multiple ascending doses
  Arms: Placebo Arm

SUMMARY:
This is a Phase 1b, multicenter, randomized, placebo-controlled, double-blind, multiple ascending dose (MAD) study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of DNL628 in participants with early Alzheimer's disease (AD), defined as mild cognitive impairment, or mild AD with biomarker evidence of amyloid positivity.

ELIGIBILITY:
Key Inclusion Criteria:

* BMI of ≥18 to < 32 kg/m2 and body weight of ≥45 kg
* Have a diagnosis of probable AD dementia based on NIA AA 2011 criteria, including amnestic or nonamnestic presentation at screening
* Have supportive evidence of AD pathology via historical records or laboratory testing at screening for amyloid positivity
* Have AD severity defined as the following at screening:

  * A Clinical Dementia Rating global score of 0.5 or 1
  * A Mini-Mental State Examination score of 20 to 30 (inclusive)

Key Exclusion Criteria:

* Have clinically significant neurological or cognitive disorders affecting the CNS other than AD, as determined by the investigator
* Have clinically significant psychiatric conditions
* Have any history of unstable or poorly controlled endocrine, pulmonary, cardiovascular, gastrointestinal, hepatic, hematological, or other significant medical condition that, in the opinion of the investigator, may interfere with the completion or interpretation of study assessment
* Have had a malignancy within 5 years before screening, except fully resected basal cell carcinoma or other malignancies (such as prostate cancer) at low risk of recurrence, depending on investigator and medical monitor agreement
* Have had previous anti amyloid or anti tau immunotherapy (including active immunization)

  * Note: ADAD participants who have participated in previous passive anti-amyloid immunotherapy > 6 months previously will be allowed, contingent on investigator and Sponsor agreement
* Have had previous exposure to gene therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) throughout the double-blind period | 37 weeks

SECONDARY OUTCOMES:
PK parameter: Maximum concentration (Cmax) of DNL628 in plasma | 37 weeks
PK Parameter: Time to reach maximum concentration (tmax) of DNL628 in plasma | 37 weeks
PK Parameter: Minimum concentration (Cmin) of DNL628 in plasma | 37 weeks
PK Parameter: Area under the concentration-time curve (AUC) from time zero to time of last measurable concentration (AUClast) of DNL628 in plasma | 37 weeks
PK Parameter: AUC from time 0 to the end of the dosing interval (AUCτ) of DNL628 in plasma | 37 weeks
PK Parameter: terminal elimination half-life (t1/2) of DNL628 in plasma | 37 weeks
PK Parameter: Accumulation ratio of DNL628 in plasma | 37 weeks
Change from baseline in total tau and ptau181 as measured in CSF | 25 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Denali Therapeutics

IPD SHARING:
Plan to Share IPD: No